CLINICAL TRIAL: NCT04835454
Title: Role of Piwi-protein Interacting RNA, miRNA-194 and Amino Acids in Patients With Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Magdy Mohammed, Assistant lecturer, Assiut University
Other Study IDs: pmapc
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Finding New Biomarkers That Could be Evaluated in Patients With Prostate Cancer and Clarify Their Role in Early Detection of Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: The control group consisted of healthy men with no cancer and no chronic diseases. They will be age-matched with patient group and recruited among men subjected to the routine periodic medical examination.
  Interventions: Diagnostic Test: piRNAs, miRNA-194, regucalcin and plasma aminoacids levels
- Prostate cancer group: Patients who are confirmed to have prostate cancer based on digital rectal examination (DRE), trasrectal ultrasonography and histopathological examination of biopsy tissue with no other coexisting cancers or prostate cancer treatment
  Interventions: Diagnostic Test: piRNAs, miRNA-194, regucalcin and plasma aminoacids levels
- benign prostatic hyperplasia group: Patients who are confirmed to have benign prostatic hyperplasia based on digital rectal examination (DRE), trasrectal ultrasonography and histopathological examination of biopsy tissue
  Interventions: Diagnostic Test: piRNAs, miRNA-194, regucalcin and plasma aminoacids levels

INTERVENTIONS:
Diagnostic Test: piRNAs, miRNA-194, regucalcin and plasma aminoacids levels — PIWI-interacting RNAs (piRNAs), a class of small nuclear RNA molecules, are associated with the PIWI proteins. MicroRNAs (miRNAs) are conserved small non-coding RNAs (19-22 nucleotide-long) that mediate post-transcriptional regulation of gene expression, affecting mRNA stability and translation by binding complementary sites on target mRNAs. Regucalcin (RGN) is an inhibitory protein of calcium signaling with calcium-binding properties. It plays a multifunctional role in the regulation of cell functions, including maintenance of intracellular calcium homeostasis, inhibitions of protein kinases and protein phosphatases linked to cell signaling process, suppressions of protein production and nuclear DNA and RNA synthesis.Free amino acids, in biological fluids can be a reduced invasive method associated to a high diagnostic potential. It was found that free amino acid profiles vary depending on type of cancer and its stage.

SUMMARY:
Prostate cancer is one of the most frequently diagnosed cancers and one of the main causes of death due to tumors in men . The mechanisms of its carcinogenesis have not been fully elucidated yet . Prostate tumours remain undetected or dormant for a long period of time before they progress loco-regionally or at distant sites as overt tumours. The molecular mechanism of dormancy is yet poorly understood

DETAILED DESCRIPTION:
Currently, early detection of prostate cancer involves mainly digital rectal examination (DRE) and testing of prostate-specific antigen (PSA) level in blood . However, over the years it became clear that PSA is not a specific biomarker of prostate cancer . Finding out new biomarkers is pivotal for early detection of prostate cancer, increasing the accuracy of diagnosis, and reducing the false positives in PSA testing These biomarkers include many biological compounds such as, microRNAs, small nuclear RNAs (sncRNA), proteins and metabolites .

PIWI-interacting RNAs (piRNAs), a class of sncRNA molecules, are associated with the PIWI proteins. Moreover, MicroRNAs (miRNAs) are conserved small non-coding RNAs (19-22 nucleotide-long) that mediate post-transcriptional regulation of gene expression, affecting mRNA stability and translation by binding complementary sites on target mRNAs[15]. Studies have shown that the miRNAs have critical roles in a variety of biological processes such as: cell proliferation, differentiation, apoptosis and carcinogenesis. Regucalcin (RGN) is an inhibitory protein of calcium signaling with calcium-binding properties. It plays a multifunctional role in the regulation of cell functions. Free amino acids, in biological fluids can be a reduced invasive method associated to a high diagnostic potential. It was found that free amino acid profiles vary depending on type of cancer and its stage.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are confirmed to have prostate cancer or benign prostatic hyperplasia based on digital rectal examination (DRE), trasrectal ultrasonography and histopathological examination of biopsy tissue

  * The control group consisted of healthy men with no cancer and no chronic diseases. They will be age-matched with patient group and recruited among men subjected to the routine periodic medical examination.

Exclusion Criteria:

* • Other coexisting cancers,

  * Prostate cancer treatment

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — A written consent will be obtained from all eligible ( aware) study participants. This consent will include whole information about the research subject and all men are free to join the research or not.
Study Population: Participants are from Urology Department, Assiut university. Patient medical history will be obtained in details. Clinical data will include age , history of previous diseases and any investigations were done. Data registered for every patient using constructed patient sheets
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
• To investigate the role of piRNAs, miRNA-194, regucalcin and aminoacids in prostate cancer development. and highlight their potential clinical utilities as biomarkers as well as potential targets for cancer treatment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Savir-Baruch B, Zanoni L, Schuster DM. Imaging of Prostate Cancer Using Fluciclovine. PET Clin. 2017 Apr;12(2):145-157. doi: 10.1016/j.cpet.2016.11.005. Epub 2017 Jan 23. PMID 28267449